CLINICAL TRIAL: NCT00243854
Title: Pilot Study Using Neoadjuvant Chemo-Radiotherapy and EGFR-tyrosine Kinase Inhibitor for Potentially Resectable Pancreatic Cancer
Brief Title: Pilot Study Using Neoadj Chemo-Rad & EGFR-tyrosine Kinase Inhibitor for Potentially Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0507-08 IUCRO-0130; NCT00216307 (obsolete NCT alias)
Record Dates: First submitted 2005-10-24; First posted 2005-10-25 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Resectable Pancreatic Cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Tarceva — Tarceva: 100mg/day x 2 weeks (Days 1-14) +

SUMMARY:
To determine the feasibility and toxicity of neoadjuvant hypofractioned radiotherapy concurrently with weekly gemcitabine and an EGFR tyrosine-kinase inhibitor (OSI-774, Tarceva) in the treatment of patients with resectable pancreatic cancer.

DETAILED DESCRIPTION:
To determine the feasibility and toxicity of neoadjuvant hypofractioned radiotherapy concurrently with weekly gemcitabine and an EGFR tyrosine-kinase inhibitor (OSI-774, Tarceva) in the treatment of patients with resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed adenocarcinoma of the pancreas
* resectable disease
* tumor </= 6cm diameter
* ECOG performance 0-1
* Organ system fxn: granulocytes (>/=1800/uL); plt ct >/=100K; bili</=2mg; liver enzymes <2.5ULN; crt </=1.5;
* Normal CXR
* Negative pregnancy test

Exclusion Criteria:

* metastatic disease or peritoneal seeding based on cross-sectional imaging
* previous irradiation to the planned field
* prior chemotherapy or immunotherapy
* active infection
* active PUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-11; Primary Completion 2010-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine if giving chemotherapy, radiation, and Tarceva,(EGFR-tyrosine kinase inhibitor)will have side effects that will prevent surgery following this therapy | Surgery - No later than 6 weeks from the completion of Neoadjuvant Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Higinia Cardenes, M.D., PhD, Principal Investigator — Indiana University; Gabriela Chiorean, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- See also: Indiana University Cancer Center website — http://cancer.iu.edu